CLINICAL TRIAL: NCT02563457
Title: Efficacy of Periodontal Treatment on Glycaemic Control in Diabetic Patients
Acronym: DIAPERIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08 031 08
Record Dates: First submitted 2015-06-23; First posted 2015-09-30 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2018-11

CONDITIONS: Diabetes
Keywords: diabetic patients; periodontal treatment; glycaemic control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- case (Experimental): diabetic patients who will receive periodontal treatment blood sampling
  Interventions: Other: periodontal manual treatment
- control (Experimental): diabetic patients without periodontal treatment (no periodontal treatment) blood sampling
  Interventions: Other: no periodontal manual treatment

INTERVENTIONS:
Other: periodontal manual treatment — periodontal manual treatment
  Arms: case
Other: no periodontal manual treatment — blood sampling
  Arms: control

SUMMARY:
This study will assess the efficacy of periodontal treatment in diabetic patient. Patients will be randomized in the periodontal group or in the control group. The control group will received a periodontal treatment after the study.

ELIGIBILITY:
Inclusion Criteria:

* patient suffering from a periodontitis
* patient with : 7,0% < Hemoglobin A1c < 9,5%

Exclusion Criteria:

* If an hospitalization is planned within the next 4 months
* Patient suffering from chronic infectious pathology (HIV, hepatitis C virus, hepatitis B virus, mononucleosis)
* Renal insufficiency
* Contra indication for amoxicilline or clindamycin
* Antithrombotic treatment
* Liver disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c blood level | 3 months
  efficacy of periodontal treatment on hemoglobin A1c

OTHER OUTCOMES:
fructosamine blood level | 3 weeks
  Compare the fructosamine content in blood between the 2 groups
Quality of life | 3 months
  Compare the quality of life between the 2 groups using the 36-Item Short Form Health Survey (SF36)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Sixou, MD, Principal Investigator — UH Toulouse
Locations (2):
- France (2):
  - UH Bordeaux, Bordeaux
  - UHToulouse, Toulouse

REFERENCES:
- [Result] Vergnes JN, Canceill T, Vinel A, Laurencin-Dalicieux S, Maupas-Schwalm F, Blasco-Baque V, Hanaire H, Arrive E, Rigalleau V, Nabet C, Sixou M, Gourdy P, Monsarrat P; DIAPERIO Group. The effects of periodontal treatment on diabetic patients: The DIAPERIO randomized controlled trial. J Clin Periodontol. 2018 Oct;45(10):1150-1163. doi: 10.1111/jcpe.13003. Epub 2018 Sep 14. PMID 30136741
- [Result] Vergnes JN, Arrive E, Gourdy P, Hanaire H, Rigalleau V, Gin H, Sedarat C, Dorignac G, Bou C, Sixou M, Nabet C. Periodontal treatment to improve glycaemic control in diabetic patients: study protocol of the randomized, controlled DIAPERIO trial. Trials. 2009 Aug 2;10:65. doi: 10.1186/1745-6215-10-65. PMID 19646281